CLINICAL TRIAL: NCT02564250
Title: Healthy Mother - Lifelong Health: A Longitudinal Study on Maternal Metabolism and Pregnancy Outcomes in Obese Pregnant Women
Brief Title: Maternal Metabolism and Pregnancy Outcomes in Obese Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: REK 2015/1017
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study longitudinal changes in maternal metabolism and pregnancy outcomes in obese pregnant women.

DETAILED DESCRIPTION:
We will study how normal metabolic changes of pregnancy are modified in obesity and investigate the consequences of altered fat and carbohydrate metabolism for pregnancy outcome. The results will aid our understanding of why pregnant obese women and their babies are at higher risk of complications and may highlight potential therapies to reduce these risks.

Overall aim and hypothesis:

The overall aim is to increase knowledge about the relation between obesity, metabolic profile/risk factors and pregnancy outcome in order to improve antenatal care and the health of the next generation.

We hypothesize that obese pregnant women can be differentiated into subgroups according to their metabolic risk profile and their risk of adverse pregnancy outcomes.

Specific aims:

Establish an outpatient clinic for obese pregnant women at Department of Obstetrics, Drammen, Vestre Viken HF in order to:

* Provide improved antenatal care for obese pregnant women who have increased risk of pregnancy complications by offering:

  * antenatal care according to national guidelines (Veileder i fødselshjelp 2014)
  * fetal surveillance (ultrasound)
  * planned delivery according to national and local guidelines
* Conduct an observational study in which clinical and biochemical data will be collected in order to increase knowledge on longitudinal metabolic changes in pregnancies complicated by obesity and how these relate to pregnancy outcomes

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with pregestational BMI > 35

Exclusion Criteria:

* diabetes mellitus type 1

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with prepregnancy BMI > 35
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | 3 years

SECONDARY OUTCOMES:
Longitudinal metabolic changes during pregnancy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marie Cecilie P Roland, PhD, Principal Investigator — Vestre Viken HF
Locations (1):
- Vestre Viken Hospital Trust, Drammen, Buskerud, Norway